CLINICAL TRIAL: NCT03453190
Title: Apremilast in Combination With Clobetasol Spray for the Treatment of Plaque Psoriasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington Dermatology Center (Other)
Responsible Party: Principal Investigator, Ronald Prussick, Principal Investigator, Washington Dermatology Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIRB1180837
Record Dates: First submitted 2018-02-26; First posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — apremilast; Clobetasol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Psoriasis Patients on Comb. Treatment (Other): Patients will be given Apremilast 30 mg bid and Clobetasol Spray 0.05 % bid on a tapering schedule over 16 weeks.
  Interventions: Combination Product: Apremilast and Clobetasol

INTERVENTIONS:
Combination Product: Apremilast and Clobetasol — Patients will receive apremilast and clobetasol with tapering dosages over 16 weeks.

SUMMARY:
Researchers want to find out if giving the drug Apremilast in combination with Clobetasol spray can help people clear their moderate to severe plaque psoriasis quicker than if Apremilast is used by itself.

DETAILED DESCRIPTION:
People over age 18 with moderate to severe plaque psoriasis who choose to be in the study and pass the four week screening period will visit the study center about 8 times over about 16 weeks. All participants will be given Apremilast, a pill that you take in the morning and at night, and which studies have shown may reduce inflammation and improve psoriasis symptoms. All participants will also be given Clobetasol to spray twice daily for two weeks, then once daily for two weeks, then every other day for two weeks. All drugs and study visits are at no cost to participants.

ELIGIBILITY:
Inclusion Criteria:

1. Must be in general good health (except for disease under study) as judged by the Sponsor Investigator, based on medical history, and physical examination. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
2. Females of childbearing potential (FCBP)† must have a negative pregnancy test at Screening and Baseline.

   Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or nonlatex condom not made out of natural [animal] membrane [for example, polyurethane]; plus one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide
3. Plaque psoriasis with at least 10% body surface area (BSA) involving the body with or without scalp lesions in adults aged 18 years and older.

Exclusion Criteria:

1. Other than disease under study, any clinically significant (as determined by the Sponsor Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
2. Any condition which would place the subject at unacceptable risk if he/she were to participate in the study.
3. Prior history of suicide attempt at any time in the subject's life time prior to screening or baseline, or major psychiatric illness requiring hospitalization within the last 3 years.
4. Pregnant or breast feeding.
5. Active substance abuse or a history of substance abuse within 6 months prior to Screening.
6. Malignancy or history of malignancy, except for:

   1. treated [ie, cured] basal cell or squamous cell in situ skin carcinomas;
   2. treated [ie, cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
7. Use of any investigational drug within 4 weeks prior to baseline, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).
8. Prior treatment with apremilast.
9. Concomitant use of drugs that treat psoriasis including but not limited to methotrexate, acitretin, cyclosporine within 4 weeks of baseline.
10. Adalimumab, etanercept, efalizumab, infliximab, or certolizumab pegol within 12 weeks prior to baseline.
11. Alefacept, briakinumab, ixekizumab, brodalumab or ustekinumab within 24 weeks prior to baseline.
12. Use of phototherapy within 4 weeks prior to baseline
13. Plaque-type psoriasis with BSA<10%
14. Psoriasis predominantly involving the face or folds (groin or axilla)
15. Psoriasis only of the palms/soles, pustular or other forms of psoriasis
16. Concurrent skin or systemic infection
17. History of intolerance to topical steroids or apremilast.
18. Topical therapy within 2 weeks of baseline (including but not limited to topical corticosteroids, topical retinoids or vitamin D analog preparations, tacrolimus, pimecrolimus, or anthralin/dithranol). Exceptions: Clobetasol Spray 0.05%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-25 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area Severity Index (PASI) | 16 weeks
  PASI is a measure of psoriatic disease severity

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Dermatology Center, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Menter A. Topical monotherapy with clobetasol propionate spray 0.05% in the COBRA trial. Cutis. 2007 Nov;80(5 Suppl):12-9. PMID 18154219
- [Background] Papp K, Cather JC, Rosoph L, Sofen H, Langley RG, Matheson RT, Hu C, Day RM. Efficacy of apremilast in the treatment of moderate to severe psoriasis: a randomised controlled trial. Lancet. 2012 Aug 25;380(9843):738-46. doi: 10.1016/S0140-6736(12)60642-4. Epub 2012 Jun 29. PMID 22748702
- [Background] Beutner K, Chakrabarty A, Lemke S, Yu K. An intra-individual randomized safety and efficacy comparison of clobetasol propionate 0.05% spray and its vehicle in the treatment of plaque psoriasis. J Drugs Dermatol. 2006 Apr;5(4):357-60. PMID 16673804
- [Background] Carey W, Glazer S, Gottlieb AB, Lebwohl M, Leonardi C, Menter A, Papp K, Rundle AC, Toth D. Relapse, rebound, and psoriasis adverse events: an advisory group report. J Am Acad Dermatol. 2006 Apr;54(4 Suppl 1):S171-81. doi: 10.1016/j.jaad.2005.10.029. PMID 16488339
- [Background] Gordon KB, Feldman SR, Koo JY, Menter A, Rolstad T, Krueger G. Definitions of measures of effect duration for psoriasis treatments. Arch Dermatol. 2005 Jan;141(1):82-4. doi: 10.1001/archderm.141.1.82. No abstract available. PMID 15655149
- [Background] Fredriksson T, Pettersson U. Severe psoriasis--oral therapy with a new retinoid. Dermatologica. 1978;157(4):238-44. doi: 10.1159/000250839. PMID 357213

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT03453190/Prot_SAP_000.pdf